CLINICAL TRIAL: NCT03318198
Title: The Effect of Intensive Inpatient Attending Supervision on Medical Errors, Patient Safety and Resident Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kathleen Finn, Inpatient Associate Program Director, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2015D005158
Record Dates: First submitted 2017-10-16; First posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Focus of Study is on Graduate Medical Education Supervision
Keywords: Graduate Medical Education; Attending Supervision of Residents; Patient Safety
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: We conducted a 9-month randomized, cross-over trial on an inpatient medicine teaching service where 22 faculty provided either: 1) direct supervision where attendings joined work rounds on established (previously admitted) patients or 2) standard supervision where attendings were available, but did not join work rounds. Each faculty member participated in both arms in random order. The primary safety outcome was rate of medical errors. Resident education was evaluated via a time motion study to assess resident participation on rounds and surveys to measure resident and attending educational ratings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Active Comparator): Attendings on the interventional arm attended daily work rounds with the resident teams in addition to established work rounds on the previously admitted patients on the care team.
  Interventions: Other: Enhanged Attending Supervision
- Control Arm (Placebo Comparator): Attendings crossed over to the control arm in which they did not attend work rounds with the team and only say new admissions with the resident team. This was usual care.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Enhanged Attending Supervision — Attendings were randomized at the start of the study to begin in the enhanced supervision arm where they attended resident work rounds. They then crossed over to the control arm where they did not attend work rounds. The outcomes were assessed between the two periods during which the attending participated in the study; attending work rounds vs. not attending work rounds.
  Arms: Intervention Arm
Other: Standard of Care — Attendings participated directly in new patient rounds but did not see patients previously known to the team with the residents.
  Arms: Control Arm

SUMMARY:
Randomized cross over trial investigating the effect of intensive attending supervision of residents caring for inpatients on the medical service on both patient safety and educational outcomes. Hypothesis: increased attending supervision would improve patient safety and resident education.

DETAILED DESCRIPTION:
Background While the relationship between resident work hours and patient safety has been extensively studied, little research has evaluated the role of attending supervision on patient safety and education.

Investigators conducted a 9-month randomized, cross-over trial on an inpatient medicine teaching service where 22 faculty provided either: 1) direct supervision where attendings joined work rounds on established (previously admitted) patients or 2) standard supervision where attendings were available, but did not join work rounds. Each faculty member participated in both arms in random order. The primary safety outcome was rate of medical errors. Secondary safety outcomes included deaths and transfers to the intensive care unit. Resident education was evaluated via a time motion study to assess resident participation on rounds and surveys to measure resident and attending educational ratings.

ELIGIBILITY:
Inclusion Criteria

* Teaching attending on the medicine service at Massachusetts General Hospital
* Resident physician on the medical service at Massachusetts General Hospital

Exclusion Criteria

* Faculty unable to complete both control and intervention arms of the study.
* Faculty unwilling to participate
* Residents unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Measurement of the rate of medical errors defined as preventable adverse events and near misses. Patient Safety Outcome | 9 months
  Using a previously validated protocol (PMID:24871238) to assess these outcomes, five research nurses reviewed the medical records, formal incident reports from the hospital incident-reporting system, daily pharmacy reports, pharmacy paging logs and solicited reports from nurses working on the study units and noted any adverse events or near misses. Four physician investigators, blinded to attending and intervention, classified each suspected incident as an adverse event, near miss or exclusion (an incident determined to be neither a medical error or adverse event). Physician reviewers further classified all adverse events as preventable or non-preventable. Medical Error rates are reports as number of events per 1,000 patient days
Resident Engagement on Rounds: Educational Outcome | 9 months
  Time motion study of the amount of time residents and faculty speak during rounds. Time was measured by a research assistant using a Microsoft access program embedded on an IPAD that recorded length of time. Time measurement outcomes are reported in minutes

SECONDARY OUTCOMES:
Resident and Faculty Perception of Education, Educational Outcome | 9 months
  A 20 question survey based on prior literature (PMID: 25340363) asking about resident and faculty experience with different levels of faculty supervision. The survey questions each were followed by a 5 point scale with a range from strongly agree, agree, neutral, disagree to strongly disagree. Strongly agree represents a better outcome. There were no subscales.
Deaths, Patient Safety Outcome | 9 months
  Hospital collected data on the number of medical patients who died during the study
Transfers to the Intensive Care Unit, Patient Safety Outcome | 9 months
  Hospital collected data on the number of medical patients who were transferred to the intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Finn, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No
The data and results from the study are listed to the research personnel associated with the study.

REFERENCES:
- [Background] Biondi EA, Varade WS, Garfunkel LC, Lynn JF, Craig MS, Cellini MM, Shone LP, Harris JP, Baldwin CD. Discordance between resident and faculty perceptions of resident autonomy: can self-determination theory help interpret differences and guide strategies for bridging the divide? Acad Med. 2015 Apr;90(4):462-71. doi: 10.1097/ACM.0000000000000522. PMID 25340363
- [Background] Starmer AJ, O'Toole JK, Rosenbluth G, Calaman S, Balmer D, West DC, Bale JF Jr, Yu CE, Noble EL, Tse LL, Srivastava R, Landrigan CP, Sectish TC, Spector ND; I-PASS Study Education Executive Committee. Development, implementation, and dissemination of the I-PASS handoff curriculum: A multisite educational intervention to improve patient handoffs. Acad Med. 2014 Jun;89(6):876-84. doi: 10.1097/ACM.0000000000000264. PMID 24871238
- [Derived] Finn KM, Metlay JP, Chang Y, Nagarur A, Yang S, Landrigan CP, Iyasere C. Effect of Increased Inpatient Attending Physician Supervision on Medical Errors, Patient Safety, and Resident Education: A Randomized Clinical Trial. JAMA Intern Med. 2018 Jul 1;178(7):952-959. doi: 10.1001/jamainternmed.2018.1244. PMID 29868877